CLINICAL TRIAL: NCT02943889
Title: The Role of Bone-marrow Derived Stem Cell Transplantation in Patients With Decompensated Liver Cirrhosis: Clinical Trial
Brief Title: Stem Cell Transplantation in Cirrhotic Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Abdeltawab Abdellah, Dr, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCT-LC
Record Dates: First submitted 2016-09-27; First posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Liver Cirrhosis
Keywords: Mesenchymal stem cells; Liver cirrhosis; Stem cell therapy
MeSH Terms: conditions — Liver Cirrhosis | interventions — Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stem cell transplantation (Experimental): This group will include 20 patients with liver cirrhosis, autologous bone marrow derived mesenchymal stem cells will be transplanted to them. Every patient will receive 2 million cells per Kg via portal vein once.
  Interventions: Biological: Mesenchymal stem cell transplantation
- Control group (No Intervention): This group will include 20 patients with liver cirrhosis as control group matching (stem cell group) in age, sex and child score. They will continue on the conventional therapy they already on and no stem cell transplantation will done for them.

INTERVENTIONS:
Biological: Mesenchymal stem cell transplantation — Bone marrow aspiration by clinical pathologist. Isolation, propagation and differentiation of stem cells will be done in stem cell center. After confirmation of the trans-differentiation into hepatocytes at the laboratory level, it will be infused into the portal vein under ultrasound guidance.
  Arms: Mesenchymal stem cell transplantation

SUMMARY:
Chronic liver disease end by liver cirrhosis and increases the risk of cancer development. Chronic liver disease in Egypt is recognized as a serious health problem affecting greater than (20 %) of the population, where the main cause is chronic infection.

Liver transplantation is still the standard treatment for advanced decompensated liver cirrhosis. However, this treatment is quite limited in clinical practice. Therefore there is a concerted effort around the world to develop regenerative and alternative therapies, so, stem cell-based therapies are emerging as new alternatives to liver transplantation for end-stage liver pathologies.

DETAILED DESCRIPTION:
This study aimed to transplant autologous bone marrow derived mesenchymal stem cells to the patients with liver cirrhosis to assess liver tissue regeneration, efficacy and safety of stem cell therapy and finally to establish an alternative treatment modality to liver transplantation.

Medical treatment of liver cirrhosis (the last stage of the illness) is very difficult that leads to high morbidity and mortality rate. Liver transplantation is still the most effective treatment for the patients with liver cirrhosis, However, serious problems are accompanied with liver transplantation, donor shortage, long waiting list, high cost, risk of rejection, operative complications and complications related to immunosuppressive drugs.

"stem cells" are cells in the human body that are capable to renew themselves and differentiate to a diverse range of specialized cell types and can be differentiated to specialized cells in appropriate medias in the laboratory. In recent years, advances in stem cell biology, have made the prospect of tissue regeneration a potential clinical reality, and several studies have shown the great promise that stem cells hold for therapy. mesenchymal stem cell based therapy has shown as promising tool in cirrhotic conditions as this type of cells have the ability to differentiate to different cell types including hepatocytes A series of studies have been performed to assess the application of bone marrow derived mesenchymal stem cells to promote liver regeneration and to alleviate cirrhosis. Some animal-based studies showed that stem cell transplantation could ameliorate liver fibrosis and improve liver functions followed by several clinical trials on human, in patients with advanced liver diseases, these studies demonstrated that stem cell transplantation could significantly reverse hepatic failure with only limited side effects. However, the effectiveness of this therapy in recent clinical trials is still conflicting and need further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated liver cirrhosis child class b or c

Exclusion Criteria:

* Patients with portal vein thrombosis, or
* Recent recurrent gastrointestinal bleeding, or
* Hepatocellular carcinoma (HCC), or
* Spontaneous bacterial peritonitis
* Pregnant or lactating women
* Vital organs failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Improvement of liver function in form of improvement in child score | 6 months

SECONDARY OUTCOMES:
Postpone or to overcome liver transplantation complications | 2 years

IPD SHARING:
Plan to Share IPD: Undecided